CLINICAL TRIAL: NCT05624320
Title: Improved Near Vision and Intermediate Without Loss of Binocular Distance Vision Using AGN-190584 in Subjects Utilizing Single -Use Daily, Contact Lenses for Distance Vision Correction in Both Eyes
Brief Title: Using AGN-190584 in Subjects Utilizing Single -Use Daily, Contact Lenses
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of interest
Sponsor: Gordon Schanzlin New Vision (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gordon Schanzlin New Vision
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2022-11

CONDITIONS: Presbyopia
Keywords: presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- single center open label, single arm study with no control and no randomization (Experimental): Investigators will enroll 30 presbyopic patients between the ages of 40-55 years old who have undergone successful contact lens fitting in single-use, daily, contact lenses between the spectacle lens powers of -4.00 -to +1.00, in both eyes for best distance correction by the primary investigator
  Interventions: Drug: AGN-190584

INTERVENTIONS:
Drug: AGN-190584 — miotic for treatment of presbyopia

SUMMARY:
AGN-190584 has gone through many clinical trials showing its safety and effectiveness in individuals from 40-55 years of age. There has been no published data on the use of this product in individuals corrected with contact lenses for distance vision. There are many other applications AGN-190584 could be used for and further studies will show the effectiveness for each.

DETAILED DESCRIPTION:
The study is a single center open label, single arm study with no control and no randomization. Investigators will enroll 30 presbyopic patients between the ages of 40-55 years old who have undergone successful contact lens fitting in single-use, daily, contact lenses between the spectacle lens powers of -4.00 -to +1.00, in both eyes for best distance correction by the primary investigator. Investigators will measure change in letters read at near and intermediate vision from baseline. Subjects will be required to apply AGN-190584 drops once daily OU. Subjects will be applying the drops on their own every day including the day of visits. During treatment investigators will measure changes in letters read from baseline in intermediate and near vision at the days 7, 14 and 21. These visits will be conducted between 2 and 4 hours after instillation of AGN-190584, with 3 hours being the target time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from age 40-55
* Prescription range: -4.00 - +1.00
* Correctable to 20/25 or better for distance
* Adapted single use contact lens patients
* Subjects able to understand the consent agreement and willing to participate

Exclusion Criteria:

* Non-contact lens wearer
* Previous use of AGN-190584
* Out of age range
* Out of prescription range
* Any corneal abnormality
* Any eye pathology
* Iritis
* Know allergy to pilocarpine

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be changes from baseline in letters read at near without loss of distance acuity (defined as loss of 5 or more letters) | 30 days

SECONDARY OUTCOMES:
secondary endpoint will be changes in intermediate letters read from baseline | 30 days

IPD SHARING:
Plan to Share IPD: No